CLINICAL TRIAL: NCT05723471
Title: Impact of a Collaborative Program of Customized, Adaptive and Supervised Physical Activity on Adherence, Fitness, Quality of Life and Resilience of Newly-diagnosed Cancer Patients
Brief Title: Impact of a Collaborative Program of Physical Activity of Newly-diagnosed Cancer Patients
Acronym: PROGRESS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/21/0600
Record Dates: First submitted 2022-11-16; First posted 2023-02-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Cancer
Keywords: Adaptative physical activity; Cancer; Quality of Life
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adaptative Physical Activity (Experimental)
  Interventions: Other: Adaptative Physical Activity
- Standard Exercise (No Intervention)

INTERVENTIONS:
Other: Adaptative Physical Activity — 12 weeks of a collaborative program of customized, adaptative and supervised physical activity by sports instructor
  Arms: Adaptative Physical Activity

SUMMARY:
During the last twenty years, the cancer overall incidence has been increasing in europe and developed countries, while diagnostic and therapeutic progress have contributes to a reduction in mortality. Currently, almost 4 million people are treated or followed for cancer in France. The physical, psychological and social after-effects are significant.

Adaptated physical activity plays an important role in the rehabilitation process. Overall, meta-analyses carried-out with most frequent cancers demonstrate that physical activity practiced would allow an improvement in quality of life, tolerance to anticancer treatments and survival.

DETAILED DESCRIPTION:
This is a multicenter, two-arm parallel-group randomizes (in a 1:1 ratio), open-label, controlled intervention clinical trial of the comparison of long term adherence to physical activity between an adaptative, customized and collaborative exercise program and standard exercise prescription in patients with newly diagnosed cancer.

ELIGIBILITY:
Inclusion Criteria:

* newly-diagnosed cancer patient
* able to start a program of physical activity within the first year follow diagnosis
* performance status between 0 to 2

Exclusion Criteria:

* uncontrolled cardiovascular disease
* peripheral neuropathy grade 3-4 with risk of falling
* bone metastasis with risk of bone fracture
* platelets <100X109/L
* hemoglobin <8g/dL
* patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of physical activity session | 2 years
  improvement of long-term adhesion to physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie MOTTON, MD, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - CHRU de Nancy, Nancy, France
  - Stéphanie MOTTON, Toulouse, France

IPD SHARING:
Plan to Share IPD: No